CLINICAL TRIAL: NCT01350570
Title: Acupuncture for Functional Bowel Disease
Brief Title: Acupuncture for Patients With Diarrhea-predominant IBS or Functional Diarrhea: a Randomized Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Collaborators: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011CB5200-Fd
Record Dates: First submitted 2011-05-06; First posted 2011-05-10 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Diarrhea-predominant Irritable Bowel Syndrome; Functional Diarrhea
Keywords: acupuncture; loperamide; functional diarrhea; IBS
MeSH Terms: interventions — Acupuncture Therapy; Loperamide

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- acupuncture group 1 (Experimental): Acupoints ST25 and BL25 will be used in the group. ST25 locate at the abdomen, while BL25 locate at the back.
  Interventions: Other: acupuncture
- acupuncture group 2 (Experimental): Acupoints LI11 and ST37 will be used in this group. LI11 is located at upper limb while ST37 is located at the lower limb.
  Interventions: Other: acupuncture group2
- acupuncture group 3 (Experimental): All acupoints used in acupuncture group1 and acupuncture group2 will be used in this group.
  Interventions: Other: acupuncture group3
- Loperamide (Active Comparator): Loperamide will be used as an active comparator to the acupuncture groups.
  Interventions: Drug: Loperamide

INTERVENTIONS:
Other: acupuncture — acupuncture group1, acupoints ST25 and BL25 will be used in this trial.
  Other Names: Acupuncture at Shumu acupoints
  Arms: acupuncture group 1
Other: acupuncture group2 — Acupoints LI11 and ST37 will be used in this group. LI11 is located at upper limb while ST37 is located at the lower limb.
  Other Names: Acupuncture at He acupoints
  Arms: acupuncture group 2
Other: acupuncture group3 — All acupoints used in acupuncture group1 and group2 will be used in this group.
  Other Names: Acupuncture at Shumu and He acupoints
  Arms: acupuncture group 3
Drug: Loperamide — Loperamide will be used in this group for a dose of 2mg a time, three time a day.
  Other Names: Luopaidingan
  Arms: Loperamide

SUMMARY:
This trial is to assess the effectiveness of three types of acupuncture for patients with functional diarrhea comparing to a positive drug control.

DETAILED DESCRIPTION:
Outcome measurements:

The frequency of bowel movement; The bristol stool scale; SF-36 evaluation

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as diarrhoea-predominant irritable bowel syndrome according to Rome III criteria;
2. Age between 18 and 65 years old;
3. Did not take any medicine for bowel symptoms and attend other clinical research;
4. Have inform consent signed.

Exclusion Criteria:

1. Diarrhea caused by diseases such as infection, etc.
2. Patients can't express himself clearly or with mental diseases;
3. Tumor and other infectious diseases;
4. With other serious diseases of Cardiovascular, liver, kidney, digestive or blood system; Pregnant women or planned to be pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Average weekly stool frequency | 4th week after inclusion
  Average weekly stool frequency, change from baseline in 4 weeks

SECONDARY OUTCOMES:
Assessment score of Bristol stool scale | 4th and 8th week after inclusion
  Bristol stool scale was designed to classify the human stool into 7 categories.
  The seven types of stool are:
  Type 1: Separate hard lumps, like nuts (hard to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft Type 5: Soft blobs with clear cut edges (passed easily) Type 6: Fluffy pieces with ragged edges, a mushy stool Type 7: Watery, no solid pieces. Entirely liquid
Assessment score of SF-36 scale | 4th and 8th after inclusion
  The Short Form (36) Health Survey (SF-36) is a survey of patient health. The SF-36 is commonly used in health economics as a variable in the quality-adjusted life year calculation to determine the cost-effectiveness of a health treatment. The chinese version of SF-36 was validated and has been widely used in acupuncture studies.
Number of patients with adverse events after treatment | 4th week after inclusion
  Number of patients with adverse events after treatment will be recorded and compared among three groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Li, MD, PhD, Principal Investigator — Chengdu University of TCM
Locations (1):
- First affiliated hospital of Chengdu university of TCM, Chengdu, Sichuan, China